CLINICAL TRIAL: NCT04260659
Title: Opioid Free vs Opioid Based Anesthesia for Laparoscopic Sleeve Gastrectomy: Clinical, Randomised Study
Brief Title: Opioid Free vs Opioid Based Anesthesia for Laparoscopic Sleeve Gastrectomy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Medical University of Warsaw (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: OFA LSG
Record Dates: First submitted 2020-01-29; First posted 2020-02-07 (Actual); Last update posted 2023-03-08 (Actual); Status verified 2023-03

CONDITIONS: Obesity; Postoperative Pain; Postoperative Nausea; Postoperative Vomiting; Opioid Use
Keywords: Opioid free anesthesia; Laparoscopic sleeve gastrectomy
MeSH Terms: conditions — Obesity; Pain, Postoperative; Postoperative Nausea and Vomiting | interventions — Dexmedetomidine; Remifentanil; Ketamine; Lidocaine; Magnesium Sulfate; Fentanyl

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Opioid liberal group (Active Comparator)
  Interventions: Drug: Remifentanil [Ultiva]
- Opioid free group (Experimental)
  Interventions: Drug: Dexmedetomidine Hydrochloride [Dexdor]; Drug: Ketamine [Ketalar]; Drug: Lidocaine [Xylocaine 2%]; Drug: Magnesium Sulphate [Inj. Magnesii Sulfurici Polpharma]; Drug: Fentanyl [Fentanyl WZF]

INTERVENTIONS:
Drug: Dexmedetomidine Hydrochloride [Dexdor] — Initial dosis of dexmedetomidine 1 mcg/kg IBW iv will be administered within 10 minutes before general anesthesia induction. Following intubation infusion of 1 mcg/kg IBW / h will be initiated and continued until the end of operation.
  Arms: Opioid free group
Drug: Remifentanil [Ultiva] — Remifentanil TCI Minto Model will be used during induction in dosis 6 ng/ml and intraoperatively appropriately to maintain hemodynamical stability.
  Arms: Opioid liberal group
Drug: Ketamine [Ketalar] — Ketamine 0,5mg/kg IBW iv will be administered during induction of general anesthesia.
  Arms: Opioid free group
Drug: Lidocaine [Xylocaine 2%] — Initial dosis of lidocaine 1,5 mg/kg IBW iv will be administered within 10 minutes before general anesthesia induction. Following intubation infusion of 3 mg/kg IBW / h will be initiated and continued until the end of operation.
  Arms: Opioid free group
Drug: Magnesium Sulphate [Inj. Magnesii Sulfurici Polpharma] — Magnesium Sulphate will be administered in dosis 50 mg/kg IBW iv intraoperatively.
  Arms: Opioid free group
Drug: Fentanyl [Fentanyl WZF] — Rescue dosis of 100 mcg iv will be administered if hypertension > 140/90 mmHg or tachycardia > 120min occurs. If necessary rescue dosis may be repeated.
  Arms: Opioid free group

SUMMARY:
Opioid free anesthesia is an anesthetic technique, in which administration of multimodal analgesia and sympathicolytics provides hemodynamic stability without use of opioids. Such management may be beneficial to the obese patients undergoing laparoscopic sleeve gastrectomy. Our study aims to compare opioid free anesthesia in such patients with standard, short-acting opioid based.

DETAILED DESCRIPTION:
The study has been approved by Bioethical Committee of Medical University of Warsaw. Informed written consent will be obtained from all patients. Sample size of 60 patients has been calculated based on the Altman normogram to obtain 30% reduction of postoperative opioid consumption with significance and power of 90%.

Consenting patients scheduled for laparoscopic sleeve gastrectomy will be randomly assigned to the computer generated list to receive opioid free or standard opioid based anesthesia.

Opioid free protocol includes administration of dexmedetomidine, lidocaine, ketamine, magnesium sulphate whereas standard group will receive remifentanil TCI Minto Model.

After the end of operation all of the patient will receive oxycodone and additional doses via PCA system for postoperative analgesia.

ELIGIBILITY:
Inclusion Criteria:

* Sleeve gastrectomy in patients with BMI > 40 or >35 with comorbidities
* Written informed consent

Exclusion Criteria:

* Patient's refusal
* Known allergies to study medication
* Inability to comprehend or participate In pain scoring scale
* Inability to use intravenous patient controlled analgesia
* Changes of operation extent during procedure
* Revisional operations

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2020-02-04 (Actual); Primary Completion 2022-10-06 (Actual); Study Completion 2023-02-22 (Actual)

PRIMARY OUTCOMES:
Total postoperative oxycodone consumption | Day "0"
  PCA (Patient's controlled analgesia) iv pump, oxycodone will be administered on patient's demand by 2mg boli, with lock out time 10 minutes
Postoperative pain score in NRS scale | Day "0", assessed 1 hour after operation
  NRS range from 0 for no pain to 10 for worst pain imaginable
Postoperative pain score in NRS scale | Day "0", assessed 6 hours after operation
  NRS range from 0 for no pain to 10 for worst pain imaginable
Postoperative pain score in NRS scale | Day "0", assessed 12 hours after operation
  NRS range from 0 for no pain to 10 for worst pain imaginable
Postoperative pain score in NRS scale | Day "1" assessed 24 hours after operation
  NRS range from 0 for no pain to 10 for worst pain imaginable

SECONDARY OUTCOMES:
Postoperative sedation score | Day "0", assessed 1,6,12 and 24 hours after operation
  1-6 Ramsay sedation score; 1 - agitated or restless 6 - unresponsive
Postoperative nausea and vomiting | Day "0", assessed 1,6,12 and 24 hours after operation
  Simplified PONV impact scale 0-6 0 - no nausea nor vomiting 6 - >3 episodes of vomiting and nausea all of the time
Rescue fentanyl administration dosis | intraoperative
  In opioid free group, rescue fentanyl dosis will be administered if hypertension > 140/90 mmHg or tachycardia > 120/min occurs
Highest BP | intraoperative
  Highest BP during operation
Lowest BP | intraoperative
  Lowest BP during operation
Highest HR | intraoperative
  Highest HR during operation
Lowest HR | intraoperative
  Lowest HR during operation
Total ephedrine dosis | intraoperative
  Ephedrine is a vasopressor used in case of hypotension to maintain mean arterial pressure > 65 mmHg or to increase blood pressure to check surgical hemostasis
Postoperative desaturation | Day "0", assessed 1,6,12 and 24 hours after operation
  SpO2 < 94%
Patient's comfort assessed in QoR-40 formulary | 7 days postoperatively
  QoR-40 scale is used to measure the quality of recovery after surgery and anesthesia, it is a 40 item questionnaire that provides a score across five dimensions: patient support, comfort, emotions, physical independence, and pain. Formulary will assess first 24 hours following the operation and will be filled by the patient 7 days after operation

CONTACTS AND LOCATIONS:
Overall Officials: Piotr Mieszczański, MD, Principal Investigator — Medical University of Warsaw
Locations (1):
- Szpital Kliniczny Dzieciatka Jezus, Warsaw, Poland

IPD SHARING:
Plan to Share IPD: Yes